CLINICAL TRIAL: NCT00960622
Title: Effect of Substituting Truvada for Combivir or Trizivir vs Continuing Combivir or Trizivir on Physiologic Correlates of Mitochondrial Function in Subjects Infected With Human Immunodeficiency Virus on Highly Active Antiretroviral Therapy
Brief Title: Switch From Combivir or Trizivir to Truvada - Mitochondrial Effects
Acronym: TRU
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: St. Luke's-Roosevelt Hospital Center (Other)
Collaborators: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TRU
Record Dates: First submitted 2009-08-17; First posted 2009-08-18 (Estimated); Results first posted 2013-03-04 (Estimated); Last update posted 2013-03-04 (Estimated); Status verified 2012-09

CONDITIONS: HIV
Keywords: treatment experienced
MeSH Terms: interventions — Emtricitabine, Tenofovir Disoproxil Fumarate Drug Combination; Emtricitabine; Tenofovir; lamivudine, zidovudine drug combination; Zidovudine; Lamivudine; abacavir, lamivudine, and zidovudine drug combination; abacavir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Truvada (Experimental): Truvada (tenofovir 300mg / emtricitabine 200mg) capsule once daily for 6 months
  Interventions: Drug: Truvada
- Combivir or Trizivir (Active Comparator): Continue on Combivir (150 mg of lamivudine, 300 mg of zidovudine) two tablets daily for 6 months or Continue on Trizivir (300 mg of abacavir as abacavir sulfate, 150 mg of lamivudine, and 300 mg of zidovudine)
  Interventions: Drug: Combivir; Drug: Trizivir

INTERVENTIONS:
Drug: Truvada — Truvada (tenofovir 300mg / emtricitabine 200mg) capsule once daily for 6 months
  Other Names: emtricitabine and tenofovir disoproxil fumarate
  Arms: Truvada
Drug: Combivir — Continue on Combivir (150 mg of lamivudine, 300 mg of zidovudine) two tablets daily for 6 months
  Other Names: Retrovir; zidovudine; Epivir; lamivudine
  Arms: Combivir or Trizivir
Drug: Trizivir — Continue on Trizivir (300 mg of abacavir as abacavir sulfate, 150 mg of lamivudine, and 300 mg of zidovudine)
  Other Names: abacavir; abacavir sulfate; lamivudine; zidovudine
  Arms: Combivir or Trizivir

SUMMARY:
Study subjects receiving the antiretroviral drugs Combivir or trizivir, will be randomized to switch to Truvada-containing highly active antiretroviral therapy (HAART) or to continue on Combivir or on trizivir. Measurements will be performed at baseline and after 6 months after randomization to either continuing on trizivir or combivir, or to switching to Truvada. Measurements include maximal or peak oxygen consumption, lactate production and clearance, subcutaneous adipose tissue and limb fat contents, insulin resistance, liver and muscle fat contents, and plasma free fatty acid concentrations. The hypothesis underlying this study is that chronic therapy with thymidine analogue nucleoside reverse transcriptase inhibitors (NRTIs), including zidovudine (AZT), leads to clinically detectable mitochondrial dysfunction in several organ systems.

DETAILED DESCRIPTION:
None different from the summary description above.

ELIGIBILITY:
Inclusion Criteria:

* infection with human immunodeficiency virus (HIV) with undetectable viral load
* on Combivir or trizivir
* able to exercise and sign consent

Exclusion Criteria:

* other active illness
* contraindication to magnetic resonance imaging (MRI) scanning or maximal exercise.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2006-08; Primary Completion 2009-07 (Actual); Study Completion 2009-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Donald P Kotler, MD, Principal Investigator — St Luke's Roosevelt Hospital New York City; Gabriel Ionescu, MD, Principal Investigator — SLRHC
Locations (1):
- St. Luke's-Roosevelt Hospital Center, New York, New York, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited from clinics.
Pre-assignment Details: Subjects had to take combivir or trizivir for at least 6 months prior to enrollment
Groups:
- Truvada 200/300 mg, Daily, by Mouth.: The study subjects will be randomly assigned to switch from Combivir or from trizivir to open-label Truvada.
- Combivir 150/300 mg, or Trizivir 300/150/300 mg Daily.: The study subjects will be randomly assigned to continue on Combivir or trizivir.This will serve as comparator group.
Period: Overall Study
Arm/Group | Truvada 200/300 mg, Daily, by Mouth. | Combivir 150/300 mg, or Trizivir 300/150/300 mg Daily.
Started | 10 | 10
Completed | 10 | 7
Not Completed | 0 | 3

BASELINE CHARACTERISTICS:
Groups:
- Truvada: switch from Combivir to Truvada
- Combivir, Trizivir.: continue on Combivir, trizivir.
- Total: Total of all reporting groups
Arm/Group | Truvada | Combivir, Trizivir. | Total
Number analyzed (Participants) | 10 | 10 | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 10 | 10 | 20
  >=65 years | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 52 (6) | 53 (4) | 53 (7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 2
  Male | 9 | 9 | 18
Region of Enrollment [Number; unit: participants]
  United States | 10 | 10 | 20

OUTCOME MEASURES:

1. Primary Outcome: Change in Peak Oxygen Uptake.
Description: change or difference in peak oxygen uptake after switching from zidovudine-based therapy, such as combivir or trizivir, to tenofovir, versus continuing on zidovudine-based therapy.The difference in peak oxygen uptake were calculated by subtracting peak oxygen uptake values at baseline from the peak oxygen uptake values after 6 months of study intervention. The changes were analyzed within each group and between groups.
Time Frame: baseline and 6 months
Measure: Mean (Standard Deviation); unit: ml/Kg/min
Groups:
- Truvada 200/300 mg, Daily, by Mouth.: switch from Combivir or trizivir to Truvada 200/300 mg, daily, by mouth.
- Combivir 150/300 mg, or Trizivir 300/150/300 mg Daily.: continue on Combivir 150/300 mg, or trizivir 300/150/300 mg daily.
Arm/Group | Truvada 200/300 mg, Daily, by Mouth. | Combivir 150/300 mg, or Trizivir 300/150/300 mg Daily.
Number analyzed (Participants) | 10 | 10
ml/Kg/min | 2.2 (8.5) | 2.8 (3.3)
Statistical Analysis 1: Comparison: Truvada 200/300 mg, Daily, by Mouth. vs Combivir 150/300 mg, or Trizivir 300/150/300 mg Daily; Paired t-tests for inter-group differences between baseline and end-of-study measurements.Regression analysis, physiological correlates of statistically significant between-group changes. P<0.05 chosen for statistical significance; Test type: Superiority or Other; p < 0.05, t-test, 2 sided; Mean Difference (Net) = 0.6, 95% CI 2-sided [-6.3 to 11.3], Standard Deviation 8.5

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Truvada | Combivir, Trizivir.
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No